CLINICAL TRIAL: NCT05874596
Title: Whole-process Quality Improvement of Patients With Acute Ischemic Stroke Undergoing Endovascular Treatment Based on an Artificial Intelligence-aided Clinical Feedback System
Brief Title: Whole-process Quality Improvement of Endovascular Treatment Basd on an AI-aided Clinical Feedback System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPTIMAL
Record Dates: First submitted 2023-05-02; First posted 2023-05-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2023-07

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): AI-aided clinical feedback system coupled with multi-aspect intervention based on the Behaviour Change Wheel model
  Interventions: Behavioral: AI-aided clinical feedback system coupled with multi-aspect intervention basd on Behaviour Change Wheel model
- Control (No Intervention): AI-aided clinical feedback system only

INTERVENTIONS:
Behavioral: AI-aided clinical feedback system coupled with multi-aspect intervention basd on Behaviour Change Wheel model — Interventions are developed on a psychological model, the Behaviour Change Wheel (BCW) .The fundamental of BCW consists of three essential elements: capability, motivation, and opportunity. Improving individual's capability, providing motivation, and increasing opportunities are goals of behaviour change intervention. To achieve the goals, 9 intervention components have been proposed in the BCW framework, and 6 components will be used in current study.
  Arms: Intervention

SUMMARY:
A clustered randomized control trial to evaluate whether multi-aspect intervention based on an AI-aided clinical feedback system could improve the quality of EVT and functional outcome of patients.

DETAILED DESCRIPTION:
Endovascular treatment (EVT) is the standard treatment for acute ischemic stroke (AIS) caused by large vessel occlusion (LVO) according to current guidelines. However, while a rapidly-growing number of stroke centers become capable of performing EVT, the general quality of EVT remains unsatisfied, resulting in a considerable proportion of patients who could not reach functional independence. Our pre-established artificial intelligence (AI)-aided clinical feedback system could dynamically record and report key timepoints of EVT in-hospital process. Combined with multi-aspect intervention via remote/on-site surveillance and education, this may be a potential solution for quality improvement of EVT. Therefore, the aim of the study is to evaluate whether an AI-aided clinical feedback system coupled with multi-aspect intervention could improve the quality of EVT. Twenty hospitals with annual EVT cases > 30 will be 1:1 randomized into intervention group and control group. The intervention group will receive AI-based clinical feedback system coupled with multi-aspect intervention, including remote/on-site surveillance and education regarding in-hospital workflow and surgical procedures of EVT. The control group only deploys AI-aided clinical feedback system. The primary outcome is the ratio of good functional outcome at 3 month.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* AIS patients receiving EVT within 24 hours of stroke onset
* Written informed consent is obtained

Exclusion Criteria:

* Patients refuse to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1289 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
Ratio of favorable functional outcome at 3 month | 3 months
  Ratio of patients with mRS ≤ 3 at 3-month follow up

SECONDARY OUTCOMES:
Ratio of good functional outcome at 3 month | 3 months
  Ratio of patients with mRS ≤2 at 3-month follow up
mRS score at 3 month | 3 months
  mRS score at 3-month follow up
Mortality at 3 month | 3 months
  Mortality at 3-month follow up
Ratio of hemorrhagic transformation at 24 hour | 24 hours
  Ratio of hemorrhagic transformation at 24 hour after EVT
Ratio of symptomatic intracranial hemorrhage at 24 hour | 24 hours
  Ratio of symptomatic intracranial hemorrhage at 24 hour after EVT
Door to groin puncture time | 24 hours
  Time interval between admission and groin puncture
Ratio of door to groin puncture time < 90 min | 24 hours
  Time interval between admission and groin puncture <90 min
Ratio of door to groin puncture time < 60 min | 24 hours
  Time interval between admission and groin puncture <60 min
Procedural duration | 24 hours
  Time interval between groin puncture and last time of digital subtraction angiography
Ratio of successful reperfusion | 24 hours
  Ratio of patients achieving modified thrombolysis in cerebral infarction (mTICI) 2b or 3

OTHER OUTCOMES:
Ratio of favorable functional outcome at 3 month in patients within 6 hours of stroke onset | 3 months
  Ratio of mRS > 2 at 3 month follow-up in patients within 6 hours of stroke onset
Door to groin puncture time in patients within 6 hours of stroke onset | 24 hours
  Time interval between admission and groin puncture in patients within 6 hours of stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Zexin Chen, Principal Investigator — Ethics committee the second affiliated hospital, school of medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No